CLINICAL TRIAL: NCT02211196
Title: Implementing Evidence-Based Tobacco Cessation Strategies in Oncology Clinics
Brief Title: Evidence-Based Tobacco Cessation Strategies in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00021885; NCI-2014-01572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU #99413 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (smoking cessation intervention) (Experimental): Participants complete a survey over approximately 10-15 minutes related to their provider's cessation advice and assistance with quitting.
  Interventions: Behavioral: smoking cessation intervention; Other: survey administration; Other: questionnaire administration

INTERVENTIONS:
Behavioral: smoking cessation intervention — Receive evidence-based tobacco cessation strategies
Other: survey administration — Ancillary studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies evidence-based tobacco cessation strategies in patients with cancer. Stop-smoking plans suggested by doctors may help patients with cancer quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess oncology providers' self-reported need for training on evidence-based tobacco cessation strategies and assess their level of interest in future training on evidence-based tobacco cessation strategies.

II. To test the feasibility of the implementation of evidence-based tobacco cessation strategies in community oncology clinics.

III. To test the feasibility of surveying community oncology patients after a clinic visit to assess provider behavior regarding screening and brief intervention for tobacco use.

OUTLINE:

Patients complete a survey over approximately 10-15 minutes related to their provider's cessation advice and assistance with quitting.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* All patients with cancer who saw a provider will be eligible

Exclusion Criteria:

* Having a nurse or lab visit only

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of providers from the Piedmont Oncology Association (POA) reporting a need for training on evidence-based tobacco cessation strategies | Up to 1 month
  Will be estimated and 95% confidence intervals (CI) constructed.
Percentage reporting feeling very confident in their ability to counsel smokers | Up to 1 month
  Will be estimated and 95% CI constructed.
Percentage reporting they would be willing to participate in training on evidence-based tobacco cessation strategies | Up to 1 month
  Will be estimated and 95% CI constructed.
Proportion of oncology patients willing to complete a survey in an oncology clinic | Up to 1 month
  Will be estimated and 95% CI constructed.
Proportion of patients who report that their provider asked about tobacco use during their visit | Up to 1 month
  These prevalences will be estimated at pre- and post-intervention, and 95% CIs calculated adjusting for the expected within-clinic correlation of patient outcomes. These outcomes will be analyzed further using a subject-specific modeling approach to account for the correlation that occurs due to patients being clustered within clinics.
Proportion of current smokers who report that their provider advised them to quit during their visit and provided tobacco-cessation strategies | Up to 1 month
  These prevalences will be estimated at pre- and post-intervention, and 95% CIs calculated adjusting for the expected within-clinic correlation of patient outcomes. These outcomes will be analyzed further using a subject-specific modeling approach to account for the correlation that occurs due to patients being clustered within clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Sutfin, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States